CLINICAL TRIAL: NCT06990633
Title: LYNX STUDY: Lynch Syndrome in Colorectal Cancer Surgery - A Multicentre, Prospective Cohort Study
Brief Title: Lynch Syndrome in Colorectal Cancer Surgery
Acronym: LYNX
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, SAADET KOCA, md ftbs phd-c, Izmir Ataturk Training and Research Hospital
Other Study IDs: Hilal
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-02

CONDITIONS: Colo-rectal Cancer; Hereditary Diseases; Lynch Syndrome
Keywords: Lynch Syndrom, Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Genetic Diseases, Inborn; Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Types of Specimens:
  Formalin-fixed, paraffin-embedded (FFPE) tumor tissue obtained from surgical resection.
  Peripheral blood samples for germline DNA extraction.
  Time of Collection:
  Tumor tissue will be collected intraoperatively.
  Blood samples will be collected postoperatively at the time of referral for genetic testing.
  Purpose of Analysis:
  Tumor tissue will undergo IHC for MMR protein expression.
  Based on IHC results, additional analyses may include BRAF mutation and MLH1 promoter methylation.
  Blood-derived germline DNA will be analyzed via next-generation sequencing (NGS) to detect pathogenic variants associated with Lynch syndrome.
  Storage and Handling:
  FFPE blocks will be stored in hospital pathology units.
  Blood samples for DNA extraction will be processed and stored according to standard protocols in certified genetic laboratories.
  Location:
  Specimens will be collected from multiple surgical centers across Türkiye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dmmr: dmmr
  Interventions: Diagnostic Test: diagnostic test
- mmr expression normal: mmr expression normal

INTERVENTIONS:
Diagnostic Test: diagnostic test — Group 1: MMR-Proficient Group Label: MMR-Proficient
  Description: Patients with normal expression of MMR proteins on IHC analysis. No indication for further genetic testing.
  Type: Observational Group
  Group 2: dMMR Group Label: dMMR
  Description: Patients with loss of MMR protein expression (MLH1, PMS2, MSH2, or MSH6) on IHC. These patients will undergo further molecular or genetic analysis to evaluate for Lynch syndrome.
  Type: Observational Group
  Groups: dmmr

SUMMARY:
Study Design (Material and Methods)

This is a multicentre, prospective cohort and audit study conducted in Türkiye. The study aims to evaluate the incidence of Lynch syndrome among patients who undergo surgery for colorectal cancer in participating general surgery departments.

Over a 12-month period, patients undergoing surgery for histologically confirmed colorectal cancer at multiple tertiary hospitals across Türkiye will be enrolled. Postoperative pathological assessments will include immunohistochemical (IHC) analysis for mismatch repair (MMR) protein expression (MLH1, PMS2, MSH2, and MSH6).

In cases showing loss of MLH1 and PMS2 expression, BRAF mutation testing will be performed. If BRAF mutation is detected, MLH1 promoter methylation analysis will follow. A positive result in both tests will suggest a sporadic etiology, whereas the absence of both findings will lead to referral for germline genetic testing using next-generation sequencing (NGS) to investigate Lynch syndrome.

For patients with isolated MSH2 and/or MSH6 loss, direct referral to genetic testing will be carried out without BRAF or methylation testing.

Patients with intact MMR expression will be recorded as the MMR-proficient control group. Comparative analysis will be conducted between dMMR and MMR-proficient patients, including demographic characteristics (age, sex, family history of cancer), tumor staging, anatomical location, and presence of metastases.

The primary outcome is to determine the incidence of Lynch syndrome among surgically treated colorectal cancer patients in Türkiye and to identify clinical and pathological correlations.

DETAILED DESCRIPTION:
Study Design (Material and Methods)

This is a multicentre, prospective cohort and audit study conducted in Türkiye. The study aims to evaluate the incidence of Lynch syndrome among patients who undergo surgery for colorectal cancer in participating general surgery departments.

Over a 12-month period, patients undergoing surgery for histologically confirmed colorectal cancer at multiple tertiary hospitals across Türkiye will be enrolled. Postoperative pathological assessments will include immunohistochemical (IHC) analysis for mismatch repair (MMR) protein expression (MLH1, PMS2, MSH2, and MSH6).

In cases showing loss of MLH1 and PMS2 expression, BRAF mutation testing will be performed. If BRAF mutation is detected, MLH1 promoter methylation analysis will follow. A positive result in both tests will suggest a sporadic etiology, whereas the absence of both findings will lead to referral for germline genetic testing using next-generation sequencing (NGS) to investigate Lynch syndrome.

For patients with isolated MSH2 and/or MSH6 loss, direct referral to genetic testing will be carried out without BRAF or methylation testing.

Patients with intact MMR expression will be recorded as the MMR-proficient control group. Comparative analysis will be conducted between dMMR and MMR-proficient patients, including demographic characteristics (age, sex, family history of cancer), tumor staging, anatomical location, and presence of metastases.

The primary outcome is to determine the incidence of Lynch syndrome among surgically treated colorectal cancer patients in Türkiye and to identify clinical and pathological correlations.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Histologically confirmed diagnosis of colorectal adenocarcinoma

Undergoing surgical resection at one of the participating general surgery departments

Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue for MMR analysis

Consent to participate in the study and undergo genetic testing if indicated

Exclusion Criteria:

Age below 18 years

Diagnosis other than colorectal adenocarcinoma

Incomplete or unavailable postoperative pathology results

Inadequate tissue samples for IHC analysis

Patients who decline participation in the study at any point

Patients who do not attend or refuse referral to genetic counseling after pathology results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) who undergo surgical resection for histologically confirmed colorectal adenocarcinoma at tertiary hospitals in Türkiye. Participants will include both elective and emergency surgical cases. All patients will have their tumor samples evaluated for MMR protein expression by immunohistochemistry. Patients with abnormal MMR expression will undergo further genetic testing. The population will represent a real-world surgical cohort, including both hereditary and sporadic colorectal cancer cases.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Lynch Syndrome Among Surgically Treated Colorectal Cancer Patients | Within 12 months following surgical resection and pathological assessment
  The primary outcome is to determine the incidence of Lynch syndrome in patients who undergo surgery for colorectal cancer. The diagnosis will be based on initial immunohistochemical (IHC) analysis of MMR protein expression (MLH1, PMS2, MSH2, MSH6), followed by molecular and germline testing (BRAF mutation, MLH1 promoter methylation, and next-generation sequencing) when indicated.